CLINICAL TRIAL: NCT04401150
Title: Lessening Organ Dysfunction With VITamin C - COVID
Brief Title: Lessening Organ Dysfunction With VITamin C - COVID-19
Acronym: LOVIT-COVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Lotte & John Hecht Memorial Foundation (Other)
Responsible Party: Principal Investigator, François Lamontagne, Co-Principal Investigator, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-31-2021-3741
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Vitamin C; COVID-19; Hospitalized Patients
Keywords: Vitamin C; COVID-19; Hospitalized patients; Pandemic; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the pharmacist of the participating site will be unblinded for the preparation of the study drug to be administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): Vitamin C: 50 mg/kg of weight administered intravenously every 6 hours for 96 hours (16 doses).
  Interventions: Drug: Vitamin C
- Control (Placebo Comparator): Normal saline (0.9% NaCl) or dextrose 5% in water (D5W) in a volume to match the vitamin C.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Vitamin C — Intravenous vitamin C administered in bolus doses of 50 mg/kg mixed in a 50-ml solution of either normal saline (0.9% NaCl) or dextrose 5% in water (D5W) during 30 to 60 minutes, every 6 hours for 96 hours (i.e. 200 mg/kg/day and 16 doses in total).
  Other Names: Ascorbic acid
  Arms: Vitamin C
Drug: Control — Dextrose 5% in water of normal saline (0.9% NaCL) in a volume to match vitamin C.
  Other Names: Placebo
  Arms: Control

SUMMARY:
LOVIT-COVID is a multicentre concealed-allocation parallel-group blinded randomized controlled trial to ascertain the effect of high-dose intravenous vitamin C compared to placebo on mortality or persistent organ dysfunction at 28 days in hospitalized COVID-19 patients.

DETAILED DESCRIPTION:
Background. Research suggests that vitamin C is potentially lifesaving in the intense inflammatory cascade such as that associated with COVID-19. Inflammation and oxidative stress are among the main mechanisms underlying COVID-19-associated acute hypoxemic respiratory failure. Previous evidence had also already established that a dysregulated inflammatory cascade may distinguish patients who transition from a relatively mild viral pneumonitis to acute respiratory distress syndrome and multiorgan failure. As such, adjunct immune modulation therapies may improve outcomes of COVID-19 patients who are hospitalized. Numerous preclinical studies have shown that, in addition to direct scavenging of oxygen radicals, vitamin C limits their production and restores endothelial function.

As the majority of hospitalized patients with COVID-19 are not critically ill, avoiding clinical deterioration and subsequent intensive care unit admission is a high priority. Participation in research should be offered before patients become critically ill, at which time many perceive that treatment may be too late. It is important to ensure that as many COVID-19 patients as possible are offered the opportunity to participate to research since that is generally the only means to access investigational therapies. The proposed trial will address this gap, by evaluating the efficacy of intravenous vitamin C in hospitalized patients with confirmed COVID-19.

Objectives. The overarching objective, which is identical to the objective of the parent LOVIT trial (NCT 03680274), is to determine whether intravenous vitamin C, compared to placebo, reduces morbidity and mortality in patients hospitalized with COVID-19. To ascertain the volume of distribution, clearance, and plasma concentration over a course of 96 hours of intravenous vitamin C 50 mg/kg of weight every 6 hours or matching placebo (pharmacokinetic (PK) substudy).

Methods. Patients will be randomly assigned to vitamin C (intravenous, 50 mg/kg every 6h) or placebo (0.9% NaCl or dextrose 5% in water) for 96 hours. Study personnel at the clinical sites will document the composite of death or persistent organ dysfunction at day 28. Daily assessments will occur for organ function, on days 1, 3, 7 for inflammation, infection, and endothelial injury biomarkers, at baseline for vitamin C level, and at 6 months for mortality and HRQoL. The LOVIT-COVID Trial will be conducted in Canadian and possibly international sites. For the PK substudy: Blood samples will be drawn around the 8th dose at time 0 and then after administration at times 1h, 2h, 4h and 6h (the 6h level will be immediately prior to the next dose). The PK substudy will be conducted with 100 participants in some of the participating centers.

Relevance. A growing body of evidence suggests that vitamin C, an inexpensive and readily available intervention, is potentially lifesaving in sepsis and may also be beneficial in COVID-19. LOVIT-COVID will constitute rigorous assessments of the effect of vitamin C monotherapy on patient-important outcomes. If proven effective, vitamin C could be used worldwide and drastically change outcomes in high- and low-income settings alike.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COVID-19;
* Admitted to hospital (ward or intensive care unit).

Exclusion Criteria:

* Receiving or has received vasopressors during the current hospitalization;
* More than 24 hours has elapsed since receipt of non-invasive ventilatory support (high-flow nasal cannula or continuous positive airway pressure or non-invasive ventilation) or invasive mechanical ventilation;
* Patient is expected to be discharged from the hospital in the next 24 hours;
* More than 14 days have elapsed since the commencement of hospital admission with respiratory illness;
* Known glucose-6-phosphate dehydrogenase (G6PD) deficiency;
* Known sickle cell anemia
* Pregnancy or breastfeeding;
* Known allergy to vitamin C;
* Known kidney stones within the past 1 year;
* Received any intravenous vitamin C during this hospitalization unless incorporated in parenteral nutrition;
* Expected death or withdrawal of life-sustaining treatments within 48 hours;
* Previously enrolled in this study;
* Previously enrolled in a trial for which co-enrolment is not allowed (co- enrolment to be determined case by case).

The trial has broad eligibility criteria and includes all COVID-19 patients admitted to the hospital (e.g. hospital ward or the intensive care unit) who are not receiving vasopressors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Death or persistent organ dysfunction | Both assessed at 28 days
  Number of deceased participants or with persistant organ dysfunction (dependency on mechanical ventilation, new renal replacement therapy, or vasopressors).

SECONDARY OUTCOMES:
Number of intensive care unit-free days | Assessed at 21 days
  Number of whole and part study days for which the patient is alive and not admitted to an intensive care unit
Persistent organ dysfunction-free days in ICU | Assessed at 28 days
  Number of study days in ICU without persistant organ dysfunction
Number of patients deceased at 6 months | 6 months
  Mortality at 6 months
Health related quality of life in 6-month survivors | 6 months
  Assessed by the EQ-5D-5L EuroQol questionnaire (EQ-5D-5L). The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ-5D visual analog scale (EQ VAS). The descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The patient is asked to indicate her/his health state by ticking the box next to the most appropriate statement in each of the 5 dimension. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the 5 dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ-VAS records the patient's self-rated health on a vertical visual analog scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Organ function | Days 1, 2, 3, 4, 7, 10, 14, 28
  Assessed by the Sequential Organ Failure Assessment (SOFA) score. Used to track a person's status during the stay in an intensive care unit to determine the extent of a person's organ function or rate of failure. The score is based on six different sub-scores, one each for the respiratory (PaO2/fraction of inspired oxygen FiO2) mmHg), cardiovascular (mean arterial pressure OR administration of vasopressors required), hepatic (liver bilirubin mg/dl [µmol/L]), coagulation (platelets x 103/µl), renal (kidneys creatinine (mg/dl) [µmol/L] (or urine output)), and neurological (Glasgow coma scale). The sub-score of each system ranges from 0 (best) to +4 (worst).
Global tissue dysoxia | Days 1, 3, 7
  Assessed by serum lactate concentration
Rate of inflammation | Days 1, 3, 7
  Assessed by interleukin-1 beta (IL-1ß), tumor necrosis factor-alpha (TNF-α), C-reactive protein (CRP).
Rate of infection | Days 1, 3, 7
  Assessed by procalcitonin (PCT).
Rate of endothelial injury | Days 1, 3, 7
  Assessed by thrombomodulin (TM) and angiopoietin-2 (ANG-2).
Occurrence of stage 3 acute kidney injury | Up to day 28
  Assessed by Kidney Disease: Improving Global Outcomes (KDIGO) criteria
Acute hemolysis | Up to day 28
  * clinician judgment of hemolysis, as recorded in the chart, OR
  * hemoglobin drop of at least 25 g/L within 24 hours of a dose of investigational product plus 2 of the following:
    * reticulocyte count >2 times upper limit of normal at clinical site lab;
    * haptoglobin <lower limit of normal at clinical site lab;
    * indirect (unconjugated) bilirubin >2 times upper limit of normal at clinical site lab;
    * lactate dehydrogenase (LDH) >2 times upper limit of normal at clinical site lab.
  Severe hemolysis:
  o hemoglobin <75 g/L AND at least 2 of the above criteria AND requires 2 units of packed red blood cells.
Hypoglycemia | During the time participants receive the 16 doses of the investigational product and the 7 days following the last dose.
  Core lab-validated glucose level <3.8 mmol/L
Vitamin C volume of distribution | 8th dose of vitamin C at time 0 (immediately prior to the dose) and then after administration at times 1 hour, 2 hours, 4 hours and 6 hours (Pharmacokynetic substudy).
  Assessed by chromatography-tandem mass spectrometry
Vitamin C clearance | 8th dose of vitamin C at time 0 (immediately prior to the dose) and then after administration at times 1 hour, 2 hours, 4 hours and 6 hours (Pharmacokynetic substudy).
  Assessed by chromatography-tandem mass spectrometry
Vitamin C plasma concentration | 8th dose of vitamin C at time 0 (immediately prior to the dose) and then after administration at times 1 hour, 2 hours, 4 hours and 6 hours (Pharmacokynetic substudy).
  Assessed by chromatography-tandem mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: François Lamontagne, MD, FRCPC, MSc, Principal Investigator — Université de Sherbrooke and CIUSSS de l'Estrie - CHUS; Neill K Adhikari, MDCM, FRCPC, MSc, Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto
Locations (2):
- Canada (2):
  - Research Center of the CHUS, Sherbrooke, Quebec
  - Research Centre of the CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] LOVIT-COVID Investigators, on behalf of the Canadian Critical Care Trials Group, and the REMAP-CAP Investigators; Adhikari NKJ, Hashmi M, Tirupakuzhi Vijayaraghavan BK, Haniffa R, Beane A, Webb SA, Angus DC, Gordon AC, Cook DJ, Guyatt GH, Berry LR, Lorenzi E, Mouncey PR, Au C, Pinto R, Menard J, Sprague S, Masse MH, Huang DT, Heyland DK, Nichol AD, McArthur CJ, de Man A, Al-Beidh F, Annane D, Anstey M, Arabi YM, Battista MC, Berry S, Bhimani Z, Bonten MJM, Bradbury CA, Brant EB, Brunkhorst FM, Burrell A, Buxton M, Cecconi M, Cheng AC, Cohen D, Cove ME, Day AG, Derde LPG, Detry MA, Estcourt LJ, Fagbodun EO, Fitzgerald M, Goossens H, Green C, Higgins AM, Hills TE, Horvat C, Ichihara N, Jayakumar D, Kanji S, Khoso MN, Lawler PR, Lewis RJ, Litton E, Marshall JC, McAuley DF, McGlothlin A, McGuinness SP, McQuilten ZK, McVerry BJ, Murthy S, Parke RL, Parker JC, Reyes LF, Rowan KM, Saito H, Salahuddin N, Santos MS, Saunders CT, Seymour CW, Shankar-Hari M, Tolppa T, Trapani T, Turgeon AF, Turner AM, Udy AA, van de Veerdonk FL, Zarychanski R, Lamontagne F. Intravenous Vitamin C for Patients Hospitalized With COVID-19: Two Harmonized Randomized Clinical Trials. JAMA. 2023 Nov 14;330(18):1745-1759. doi: 10.1001/jama.2023.21407. PMID 37877585